CLINICAL TRIAL: NCT00417157
Title: Successful Application of Modified Natural Cycle in Poor Responders With High Basal FSH Prior to Oocyte Donation
Brief Title: Modified Natural Cycle Offers a Chance of Pregnancy in Patients With Poor Response and High Basal FSH
Status: Completed | Type: Observational
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Other Study IDs: MNC
Record Dates: First submitted 2006-12-22; First posted 2006-12-29 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Infertility; Premature Ovarian Failure
Keywords: GnRH antagonist; Poor responders; Oocyte donation; Modified natural cycle
MeSH Terms: conditions — Infertility; Primary Ovarian Insufficiency | interventions — follitropin beta; ganirelix; Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: recombinant FSH (Puregon, Organon, The Netherlands)
Drug: GnRH antag: Ganirelix (Orgalutran, Organon, The Netherlands)
Drug: hCG (Pregnyl, Organon, The Netherlands)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a modified natural cycle in patients with previous poor response to infertility drugs and high basal FSH, prior to proceeding to oocyte donation or abandoning fertility treatment.

DETAILED DESCRIPTION:
Poor responders are a diverse group of IVF patients who fail to respond to IVF drugs. In these patients pregnancy rates remain disappointingly low and usually oocyte donation is their only viable option. The need for lengthy ovarian stimulation regimes can be avoided by performing IVF during a natural menstrual cycle. However, the main problem with a natural cycle is that successful IVF outcome can be compromised by a premature LH surge. This problem can be solved by the administration of GnRH antagonists that suppress endogenous gonadotropin levels, comprising a modified natural cycle (MNC). Previous studies have shown that MNC offers no realistic chances of pregnancy prior to oocyte donation. In this study we will re-assess this view by showing that MNC offers some, albeit small, chances of positive IVF outcome in patients with known previous poor response prior to oocyte donation.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycle (21-35 days)
* Basal FSH>12 IU/ml
* One or more failed IVF attempts (<3 oocyte retrieved)

Exclusion Criteria:

* PCOS
* Normal responders

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women undergoing IVF treatment
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Live birth per started cycle | live birth

SECONDARY OUTCOMES:
Biochemical pregnancy per started cycle | positive hCG test 14 days post oocyte retrieval
Clinical pregnancy per started cycle | presence of fetal sac and heart beat at 7 weeks of gestation
Cycle cancellation rates | cycles not reaching oocyte retrieval
Ongoing pregnancy rates per started cycle | presence of fetal sac and heart beat at 12 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon Lainas, PhD, Principal Investigator — Eugonia
Locations (1):
- Eugonia, Athens, Greece

REFERENCES:
- [Background] Kolibianakis E, Zikopoulos K, Camus M, Tournaye H, Van Steirteghem A, Devroey P. Modified natural cycle for IVF does not offer a realistic chance of parenthood in poor responders with high day 3 FSH levels, as a last resort prior to oocyte donation. Hum Reprod. 2004 Nov;19(11):2545-9. doi: 10.1093/humrep/deh452. Epub 2004 Oct 7. PMID 15471941